CLINICAL TRIAL: NCT05366257
Title: Real-world Resource Use and Costs of CAR-T Therapies in Diffuse Large B-cell Lymphoma (DLBCL): Inpatient and Outpatient Settings
Brief Title: Real-world Resource Use and Costs of CAR-T Therapies in Diffuse Large B-cell Lymphoma (DLBCL)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019CUS08
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Diffuse Large B-cell Lymphoma (DLBCL)
Keywords: CAR-T,; DLBCL,; Inpatient,; Outpatient
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CAR-T: Inpatient (IP) Cohort: Patients received CAR-T infusion in IP setting
  Interventions: Other: CAR-T
- CAR-T: Outpatient (OP) Cohort: Patients received CAR-T infusion in OP setting
  Interventions: Other: CAR-T
- Allo-HSCT cohort: Patients received allogeneic hematopoietic stem cell transplant
  Interventions: Other: Allo-HSCT cohort

INTERVENTIONS:
Other: CAR-T — infusion of CAR-T therapy among patients with r/r DLBCL
  Groups: CAR-T: Inpatient (IP) Cohort; CAR-T: Outpatient (OP) Cohort
Other: Allo-HSCT cohort — Patients received allogeneic hematopoietic stem cell transplant
  Groups: Allo-HSCT cohort

SUMMARY:
A retrospective, non-interventional cohort study was used to address the study objectives. This study aimed to provide a better understanding of real-world healthcare resource utilization (HRU) and healthcare reimbursement costs associated with CAR-T therapy among patients with r/r Diffuse Large B-cell Lymphoma (DLBCL).

DETAILED DESCRIPTION:
A retrospective, non-interventional cohort study was used to address the study objectives. This study aimed to provide a better understanding of real-world HRU and healthcare reimbursement costs associated with CAR-T therapy among patients with r/r DLBCL.

Eligible adult patients with r/r DLBCL who were treated with CAR-T therapy or allo-HSCT between January 1, 2017 to September 31, 2019 were identified from the Centers for Medicare & Medicaid Services (CMS) 100% Medicare Database. The CAR-T cohort was further classified into CAR-T IP and CAR-T OP cohorts based on the infusion setting.

The index date was defined as the date of CAR-T therapy administration or allo-HSCT. Baseline period was defined as three months prior to the index date. Study period was defined from the index date to the end of health plan coverage based on insurance enrollment file or death, whichever occurred earlier.

Two sets of comparisons on HRU and healthcare reimbursement costs were conducted, one between IP vs. OP infusion of CAR-T, and the other between patients who received CAR-T therapy vs. allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

CAR-T cohort:

* Patients had at least one International Classification of Diseases, Tenth Revision (ICD- 10) diagnosis code for DLBCL.
* Patients received CAR-T therapy following DLBCL diagnosis. The administration date of CAR-T therapy was defined as the index date. Patients who received both CAR-T therapy and allo-HSCT were classified based on the first treatment that the patient received
* Patients were at least 18 years of age as of the index date
* Patients had at least three months of continuous eligibility in the Medicare Part A and Part B data before the index date. Since 2019 Part D data is not available in the current data cut, eligibility requirement in the Part D data was not required

Patients were further classified into CAR-T IP and CAR-T OP cohorts depending on where the administration occurred.

Allo-HSCT cohort:

* Patients had at least one ICD-10 diagnosis code for DLBCL.
* Patients received allo-HSCT following DLBCL diagnosis. The date of allo-HSCT procedure was defined as the index date. Patients who received both CAR-T therapy and allo-HSCT were classified based on the first treatment the patient received
* Patients were at least 18 years of age as of the index date
* Patients had at least three months of continuous eligibility in the Medicare Part A and Part B data before the index date. Since 2019 Part D data is not available in the current data cut, eligibility requirement in the Part D data was not required

Exclusion Criteria:

- Patients had a medical claim associated with a clinical trial (ICD-9 CM code V70.7; ICD-10 CM code Z00.6) during one month before and after the index date

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with DLBCL who received CAR-T therapy or allo-HSCT procedure between January 1, 2017 to September 31, 2019
Sampling Method: Non-Probability Sample
Enrollment: 160602 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
Mean length of follow-up in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Mean length of follow up was reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of patients with IP visit in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of patients with IP visit were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of IP admissions in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of IP admissions were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of IP days in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of patients with IP visit were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of ICU stays in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of ICU stays were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of ICU days in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of ICU days were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of patients with OP visit in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of patients with OP visit were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of OP visits in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of OP visits were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of patients with ER visit in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of patients with ER visit were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Number of ER visits in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of ER visits were reported to compare Health Resource Use (HRU) between IP vs. OP infusion of CAR-T therapy among patients with r/r DLBCL.
Total healthcare reimbursement costs in CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Total healthcare reimbursement costs, including medical service costs and pharmacy costs, inflated to 2020 US dollars (USD) were reported in CAR-T IP and CAR-T OP cohorts.

SECONDARY OUTCOMES:
Mean length of follow-up for CAR-T therapy vs. allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Mean length of follow up was reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of patients with IP visit in CAR-T vs allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of patients with IP visit were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of IP admissions in CAR-T therapy vs. allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of IP admissions were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of IP days in CAR-T therapy vs. allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of IP days were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of ICU stays in CAR-T therapy vs. allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of ICU stays were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of ICU days in CAR-T therapy vs. allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of ICU days were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of patients with OP visit in CAR-T vs allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of patients with OP visit were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of OP visits in CAR-T therapy vs. allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of OP visits were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of patients with ER visit in CAR-T vs allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of patients with ER visit were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
Number of ER visits in CAR-T therapy vs. allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Number of ER visits were reported to compare Health Resource Use (HRU) of CAR-T therapy vs. allo-HSCT among patients with r/r DLBCL.
IP re-admission/admission among CAR-T IP and OP cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  IP re-admission/admission were reported to assess post-infusion IP admission/readmission among patients with r/r DLBCL who received CAR-T therapy.
AE rate during the study period among CAR-T cohorts | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Rate of adverse events (AEs) were reported among patients with r/r DLBCL who received CAR-T therapy.
Cost of AEs among CAR-T cohorts during the study period | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Cost per AE event were reported among patients with r/r DLBCL who received CAR-T therapy.
Total healthcare reimbursement costs in CAR-T vs allo-HSCT cohort | throughout the study, approximately 2 years ( January 1, 2017 to September 31, 2019)
  Total healthcare reimbursement costs, including medical service costs and pharmacy costs, defined as the amount paid by Medicare, inflated to 2020 USD were reported in overall CAR T and allo-HSCT cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CCTL019CUS08 from the Novartis Clinical Trials Results Databse — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17931